CLINICAL TRIAL: NCT05531058
Title: [AI-driven Vaccine Communicator: the Impact of a Web-based Psychoeducation Programme with a Motivational AI-based Digital Assistant on Covid-19 Vaccine Hesitancy in Hong Kong's Population
Brief Title: The Impact of a Web-based Psychoeducation Programme with a Motivational AI Chatbot on Covid-19 Vaccine Hesitancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P0039051
Record Dates: First submitted 2022-08-28; First posted 2022-09-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2022-08

CONDITIONS: Vaccine Hesitancy; COVID-19
Keywords: Vaccine Hesitancy; COVID-19; Motivational Intervention; AI Chatbot; Artificial Intelligence
MeSH Terms: conditions — Vaccination Hesitancy; COVID-19

STUDY DESIGN:
Intervention Model Description: We aim to have two study group, including the AI-driven vaccine communicator intervention group and the self-learning of COVID-19 vaccine knowledge control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI-driven vaccine communicator intervention group (Experimental): The intervention will include five modules web-based psychoeducation programme (two modules sessions weekly, each module lasts for 15-20 minutes) which includes educational materials, animations of vaccine research and development, and an MI communication skills-based AI, digital assistant.
  Interventions: Behavioral: AI-driven Vaccine Communicator
- Self-learning of COVID-19 vaccine knowledge control group (Active Comparator): Participants in the control group will be given HK government websites in COVID-19 vaccine and invite to join the online examination in relation to Covid-19 vaccine knowledge.
  Interventions: Behavioral: Self-learning of COVID-19 vaccine knowledge

INTERVENTIONS:
Behavioral: AI-driven Vaccine Communicator — The intervention will include five modules web-based psychoeducation programme (two module sessions weekly, each module lasts for 15-20 minutes) and interact with an MI communication skills-based AI, digital assistant.
  Arms: AI-driven vaccine communicator intervention group
Behavioral: Self-learning of COVID-19 vaccine knowledge — Participants in the control group will be given HK government websites in COVID-19 vaccine and invite to join the online examination in relation to Covid-19 vaccine knowledge (using multiple choices questions similar to the intervention group), and this is to ensure that participants from the control group also use time to search relevant information of covid-19 vaccines, also this is to control the time effects.
  Arms: Self-learning of COVID-19 vaccine knowledge control group

SUMMARY:
Vaccine hesitancy is defined as 'delay in acceptance or refusal of vaccines, despite the availability of vaccine service' and was named one of the top ten global health threats by the World Health Organization in 2019.

Our proposed study will aim to develop and evaluate the effectiveness of a Web-based psychoeducation programme to address Covid-19 vaccine hesitancy, 'AI-driven Vaccine Communicator' (including educational materials, animations of vaccine research and development, and an MI communication skills-based AI, digital assistant).

Our goal is to standardise our intervention so that it can serve as an effective toolkit for clinicians/healthcare providers to increase Hong Kong residents' motivation to vaccinate and to ensure that the programme can be adapted to viral mutations and newly developed vaccines in the medium/long term.

DETAILED DESCRIPTION:
This study is a two-arm, single-blind pilot randomized controlled trial, and it will be adopted to evaluate the efficacy of the 'AI-driven Vaccine Communicator' relative to being self-informed about Covid-19 vaccines.

Also, to address the widespread hesitancy among Hong Kong residents toward Covid-19 vaccines, we will develop a Web-based psychoeducation programme, 'AI-driven Vaccine Communicator,' driven by artificial intelligence (AI) techniques based on the Vaccine Hesitancy Determinants Matrix Model and MI communication skills and concepts (theoretical underpinnings). After developing and piloting this programme, we will test its effectiveness among members of the population who are hesitant about Covid-19 vaccines. The programme will then be refined further and standardised to use the most relevant information and effective communication skills to promote acceptance of Covid-19 vaccines among a wider Hong Kong population. Clinicians and healthcare providers will be able to utilise our programme as a toolkit in their usual practice when working with clients who are hesitant about Covid-19 vaccines.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or above;
* Hong Kong residents;
* Show vaccine hesitancy (not taking COVID-19 vaccines or receiving involuntary COVID-19 vaccines);
* have internet access
* able to read Chinese or English. Recruitment involved social media promotion and collaborating with community organizations

Exclusion Criteria:

* People with self-reported cognitive impairments or mental disorders that might interfere with their understanding of the intervention content;
* People who currently engaged in another clinical trial in relation to Covid-19 vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Vaccine hesitancy at pre-test | Vaccine hesitancy will be assessed at pre-intervention.
  Vaccine hesitancy measured by Adult Vaccine Hesitancy scale and a single question 'plan for next dose'
Vaccine hesitancy at post-intervention | Vaccine hesitancy will be assessed five weeks post the commencement of the intervention (at post-intervention).
  Vaccine hesitancy measured by Adult Vaccine Hesitancy scale and a single question 'plan for next dose'
Vaccine hesitancy at three months follow-up | Vaccine hesitancy will be assessed after three months follow-up.
  Vaccine hesitancy measured by Adult Vaccine Hesitancy scale and a single question 'plan for next dose'
Vaccine hesitancy at six months follow-up | Vaccine hesitancy will be assessed after six months follow-up.
  Vaccine hesitancy measured by Adult Vaccine Hesitancy scale and a single question 'plan for next dose'

SECONDARY OUTCOMES:
Vaccine confidence at pre-test | Vaccine confidence will be assessed at pre-intervention.
  Vaccine confidence assessed by Vaccine Confidence Index scale
Vaccine confidence at post-intervention | Vaccine confidence will be assessed five weeks post the commencement of the intervention (at post-intervention).
  Vaccine confidence assessed by Vaccine Confidence Index scale
Vaccine confidence at three months follow-up | Vaccine confidence will be assessed after three months follow-up.
  Vaccine confidence assessed by Vaccine Confidence Index scale
Vaccine confidence at six months follow-up | Vaccine confidence will be assessed after six months follow-up.
  Vaccine confidence assessed by Vaccine Confidence Index scale
Vaccine readiness at pre-test | Vaccine readiness will be assessed at pre-intervention.
  Participants' perception of their degree of attitudinal change using three one-item measures of readiness for vaccine perception: How important is it for you to receive a COVID-19 vaccine?; How ready are you to receive a COVID-19 vaccine?; How confident are you about receiving a COVID-19 vaccine?
Vaccine readiness at post-intervention | Vaccine readiness will be assessed five weeks post the commencement of the intervention (at post-intervention).
  Participants' perception of their degree of attitudinal change using three one-item measures of readiness for vaccine perception: How important is it for you to receive a COVID-19 vaccine?; How ready are you to receive a COVID-19 vaccine?; How confident are you about receiving a COVID-19 vaccine?
Vaccine readiness at three months follow up | Vaccine readiness will be assessed after three months follow-up.
  Participants' perception of their degree of attitudinal change using three one-item measures of readiness for vaccine perception: How important is it for you to receive a COVID-19 vaccine?; How ready are you to receive a COVID-19 vaccine?; How confident are you about receiving a COVID-19 vaccine?
Vaccine readiness at six months follow up | Vaccine readiness will be assessed after six months follow-up.
  Participants' perception of their degree of attitudinal change using three one-item measures of readiness for vaccine perception: How important is it for you to receive a COVID-19 vaccine?; How ready are you to receive a COVID-19 vaccine?; How confident are you about receiving a COVID-19 vaccine?
Vaccine-Related Health Literacy at pre-test | Vaccine-Related Health Literacy will be assessed at pre-intervention.
  Vaccine-Related Health Literacy assessed by Chinese version of the European Health Literacy Survey Questionnaire
Vaccine-Related Health Literacy at post-intervention | Vaccine-Related Health Literacy will be assessed five weeks post the commencement of the intervention (at post-intervention).
  Vaccine-Related Health Literacy assessed by Chinese version of the European Health Literacy Survey Questionnaire
Vaccine-Related Health Literacy at three months follow up | Vaccine-Related Health Literacy will be assessed after three months follow-up.
  Vaccine-Related Health Literacy assessed by Chinese version of the European Health Literacy Survey Questionnaire
Vaccine-Related Health Literacy at six months follow up | Vaccine-Related Health Literacy will be assessed after six months follow-up.
  Vaccine-Related Health Literacy assessed by Chinese version of the European Health Literacy Survey Questionnaire
Trust in government at pre-test | Trust in government will be assessed at pre-intervention.
  Trust in government will be measured with the four-item Vaccine Confidence Index.
Trust in government at post-test | Trust in government will be assessed five weeks post the commencement of the intervention (at post-intervention).
  Trust in government will be measured with the four-item Vaccine Confidence Index.
Trust in government at three-months follow up | Trust in government will be assessed after three-months follow up.
  Trust in government will be measured with the four-item Vaccine Confidence Index.
Trust in government at six-months follow up | Trust in government will be assessed after six-months follow up.
  Trust in government will be measured with the four-item Vaccine Confidence Index.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, Dr, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, The Hong Kong Polytechnic Unviersity, Hong Kong, Hong Kong

REFERENCES:
- [Background] Jarrett C, Wilson R, O'Leary M, Eckersberger E, Larson HJ; SAGE Working Group on Vaccine Hesitancy. Strategies for addressing vaccine hesitancy - A systematic review. Vaccine. 2015 Aug 14;33(34):4180-90. doi: 10.1016/j.vaccine.2015.04.040. Epub 2015 Apr 18. PMID 25896377
- [Background] MacDonald NE; SAGE Working Group on Vaccine Hesitancy. Vaccine hesitancy: Definition, scope and determinants. Vaccine. 2015 Aug 14;33(34):4161-4. doi: 10.1016/j.vaccine.2015.04.036. Epub 2015 Apr 17. PMID 25896383
- [Background] Taylor S, Landry CA, Paluszek MM, Groenewoud R, Rachor GS, Asmundson GJG. A Proactive Approach for Managing COVID-19: The Importance of Understanding the Motivational Roots of Vaccination Hesitancy for SARS-CoV2. Front Psychol. 2020 Oct 19;11:575950. doi: 10.3389/fpsyg.2020.575950. eCollection 2020. PMID 33192883
- [Background] Gagneur A, Lemaitre T, Gosselin V, Farrands A, Carrier N, Petit G, Valiquette L, De Wals P. A postpartum vaccination promotion intervention using motivational interviewing techniques improves short-term vaccine coverage: PromoVac study. BMC Public Health. 2018 Jun 28;18(1):811. doi: 10.1186/s12889-018-5724-y. PMID 29954370
- [Background] Leung SF, Ma J, Russell J. Enhancing motivation to change in eating disorders with an online self-help program. Int J Ment Health Nurs. 2013 Aug;22(4):329-39. doi: 10.1111/j.1447-0349.2012.00870.x. Epub 2012 Aug 6. PMID 22882349